CLINICAL TRIAL: NCT07216729
Title: Evaluating the Effects of Lactobacillus Reuteri DSM 17938 on State and Trait Stress in Stressed Adults
Brief Title: The Effects of Probiotic Supplementation on State and Trait Stress, Anxiety, and Depression Symptoms in Stressed Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Responsible Party: Principal Investigator, Lauren Finkelstein, Principal Investigator, University of Colorado, Boulder
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 22-0234
Record Dates: First submitted 2025-10-10; First posted 2025-10-15 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Anxiety Symptoms; Perceived Stress; Depressive Symptoms
Keywords: Lactobacillus reuteri DSM 17938; Perceived stress; Anxiety; Depression; Probiotic; Randomized controlled trial
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): 5 drops daily (100 million colony-forming units) for 46 days of Lactobacillus reuteri DSM 17938 in sunflower oil, medium chain triglyceride oil, and silicon dioxide.
  Interventions: Dietary Supplement: Lactobacillus reuteri DSM 17938
- Placebo (Placebo Comparator): 5 drops daily for 46 days of a placebo consisting of the inactive ingredients from the probiotic supplement, specifically sunflower oil, medium chain triglyceride oil, and silicon dioxide.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus reuteri DSM 17938 — 5 drops (100 million CFUs) daily for 46 days of L. reuteri DSM 17938 in sunflower oil, medium chain triglyceride oil, and silicon dioxide.
  Arms: Probiotic
Other: Placebo — 5 drops daily for 46 days of placebo consisting of inactive ingredients from probiotic supplement, specifically sunflower oil, medium chain triglyceride oil, and silicon dioxide.
  Arms: Placebo

SUMMARY:
The goal of this randomized controlled trial is to learn if supplementation with the probiotic Lactobacillus reuteri DSM 17938 can reduce levels of trait and state perceived stress, anxiety, and depressive symptoms compared to a placebo in a population of stressed adults ages 18-45. This study also investigates several evidence-based moderators of treatment effects, evaluates whether the probiotic caused side effects, and evaluates whether effects endured at 1-month post-supplementation.

ELIGIBILITY:
Inclusion Criteria:

* age 18 - 45
* scoring 14+ on the perceived stress scale-10 indicating medium stress or higher
* ability to provide informed consent
* willingness not to take probiotic supplements (pills, tablets, oils, etc.) other than the product provided in the clinical study until all study procedures are completed
* own a smartphone and are willing to receive study materials and complete study procedures by text

Exclusion Criteria:

* a history of gastrointestinal discomfort or surgery, urinary incontinence, cancer, toxic shock syndrome, frequent diarrhea, vital signs outside of the acceptable range (i.e., blood pressure >160/100, oral temperature >100°F, pulse >100), heart disease, heart attack, lung/respiratory disease, any pulmonary, cardiovascular, gastrointestinal, hepatic or renal functional abnormality (i.e. a medical diagnosis related to lungs, heart, stomach/intestines, liver, or kidneys), HIV, Hepatitis B, Hepatitis C, bipolar disorder, psychosis, or confirmed or suspected immunosuppression or immunodeficiency
* current (past month) alcohol or substance abuse or dependence (score of 2+ on the UNCOPE)
* consistent (e.g., 5x/week or greater) probiotic supplementation within the last month, including probiotic food products such as yogurt
* receiving antibiotics within the last month
* receiving medications that interfere with gut motility (opiates, loperamide, stool softeners)
* use of systemic antibiotics, antifungals, antivirals, or antiparasitics (intravenous, intramuscular, or oral)
* use of oral, intravenous, intramuscular, nasal or inhaled corticosteroids
* use of cytokines or cytokine inhibitors
* use of methotrexate or immunosuppressive cytotoxic agents
* receiving immunosuppressive drugs/medications or treatment including antineoplastic therapy, post-transplantation immunosuppressive therapy, and/or radiation therapy
* participation in conflicting interventional research protocol
* unstable dietary history as defined by major changes in diet during the previous month, where the subject has eliminated or significantly increased a major food group in their diet
* female who is pregnant or lactating or reports expecting to get pregnant during the course of the study
* currently involved in the criminal justice system as a prisoner or ward of the state

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2024-05-06 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean trait perceived stress as assessed by PSS-10 | Baseline and the end of treatment at 46 days
  Perceived stress scale-10 (PSS-10) administered via REDCap. Possible score range of 0 to 40, with 0-13 considered low stress, 14-26 moderate stress, and 27-40 high stress.
State perceived stress as assessed by adapted PSS-4 using ecological momentary assessment | Five times per day (hourly, 12-7pm, sent via text with a 15 minute response window) during the last 5 days of supplementation, days 42 to 46, when the investigators expect participants to have reached maximum benefit
  Perceived stress scale-4 (PSS-4) administered via REDCap and adapted for state measurement. The investigators adapted this measure for state stress by asking participants to rate the intensity of perceived stress they were experiencing in the moment, as opposed to the frequency with which they experienced perceived stress over the past month. Possible score range of 0 to 16, with higher scores indicating higher levels of state stress.

SECONDARY OUTCOMES:
Change from baseline in mean trait anxiety symptoms as assessed by GAD-7 | Baseline and the end of treatment at 46 days
  Generalized Anxiety Disorder-7 scale (GAD-7) administered via REDCap. Possible score range of 0 to 21, with higher scores indicating higher levels of anxiety symptoms.
State anxiety symptoms as assessed with the SUDS using ecological momentary assessment | Five times per day (hourly, 12-7pm, sent via text with a 15 minute response window) during the last 5 days of supplementation, days 42 to 46, when the investigators expect participants to have reached maximum benefit
  Subjective units of distress scale (SUDS) administered via REDCap. Possible score range of 0 to 100, with higher scores indicating higher levels of state anxiety.
Change from baseline in mean trait depressive symptoms as assessed by the PHQ-8 | Baseline and the end of treatment at 46 days
  Patient Health Questionnaire-8 (PHQ-8) administered via REDCap. Possible score range of 0 to 24, with higher scores indicating higher levels of depression.
State depressive symptoms as assessed by SUDS using ecological momentary assessment | Five times per day (hourly, 12-7pm, sent via text with a 15 minute response window) during the last 5 days of supplementation, days 42 to 46, when the investigators expect participants to have reached maximum benefit
  Subjective Units of Distress Scale (SUDS) administered via REDCap. Possible score range of 0 to 100, with higher scores indicating higher levels of state depression.

OTHER OUTCOMES:
Side effects as assessed on the final day of supplementation using the GASE | End of treatment at day 46
  Generic Assessment of Side Effects (GASE), excluding the question assessing suicidality and administered on REDCap. This measure assesses 35 of the most common subjective side effects of clinical trials (e.g., nausea), and asks participants to rate whether they experienced each complaint on a scale from 0 ("not present") to 3 ("severe"). If they endorsed experiencing a side effect (score of 1+), participants were then asked whether the complaint related to the probiotic (yes/no).

CONTACTS AND LOCATIONS:
Overall Officials: Lauren B Finkelstein, MA, Principal Investigator — University of Colorado, Boulder
Locations (1):
- University of Colorado Boulder, Muenzinger Psychology Building, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data (IPD) will be shared with other researchers in our lab to conduct secondary analyses. Data sharing will ensure protection of participant confidentiality.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning late summer/early fall of 2024 with no end date
Access Criteria: Faculty advisor who oversaw the initial trial is supervising another graduate student to use the data to address research questions outlined in the IRB-approved protocol, in addition to some secondary analyses.

REFERENCES:
- See also: Prior pre-registration on Open Science Framework, initially submitted prior to starting data collection — https://osf.io/a6htn